CLINICAL TRIAL: NCT02857218
Title: A Pilot Study Using a Novel Imaging of Lymph Nodes in Patients With Locally Advanced Esophageal Cancer Using Ferumoxytol Enhanced MRI
Brief Title: Ferumoxytol-Enhanced MRI in Imaging Lymph Nodes in Patients With Stage IIB-IIIC Esophageal Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alexander Guimaraes, Associate Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00012071; NCI-2016-01093 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00012071 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Stage IIB Esophageal Cancer AJCC v7; Stage III Esophageal Cancer AJCC v7; Stage IIIA Esophageal Cancer AJCC v7; Stage IIIB Esophageal Cancer AJCC v7; Stage IIIC Esophageal Cancer AJCC v7
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (ferumoxytol, MRI) (Experimental): Patients receive ferumoxytol IV over 15 minutes and then undergo ferumoxytol-enhanced MRI (Magnetic Resonance Imaging) after 24-36 hours and before surgery at week 12.
  Interventions: Drug: Ferumoxytol; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol — Undergo ferumoxytol-enhanced MRI
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Procedure: Magnetic Resonance Imaging — Undergo ferumoxytol-enhanced MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This pilot clinical trial studies how well ferumoxytol-enhanced magnetic resonance imaging (MRI) works in imaging lymph nodes in patients with stage IIB-IIIC esophageal cancer. Ferumoxytol is a form of very small iron particles that are taken up by cells in normal lymph nodes and may work better in imaging patients with esophageal cancer when paired with MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine feasibility of administering ferumoxytol and obtaining ferumoxytol enhanced magnetic resonance (MR) images in patients with resectable locally advanced esophageal cancer before starting neoadjuvant chemoradiation therapy and again before esophagectomy.

SECONDARY OBJECTIVES:

I. To collect detailed information about the location of ultrasmall superparamagnetic iron oxide (USPIO)-MRI detected lymph nodes prior to neoadjuvant chemoradiation therapy and again prior to esophagectomy.

II. To determine the sensitivity and specificity of ferumoxytol enhanced MR imaging in the assessment of pathologic lymph node involvement based on pathological findings at the time of esophagectomy.

OUTLINE:

Patients receive ferumoxytol intravenously (IV) over 15 minutes and then undergo ferumoxytol-enhanced MRI after 24-36 hours and before surgery at week 12.

After completion of study treatment, patients are followed up for 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, locally advanced, malignancy of the esophagus; the cancer may involve the stomach up to 5 cm; based on multi-disciplinary tumor board discussion, patients are candidates for tri-modality treatment
* Stage T1-4aN1-2, by the American Joint Committee on Cancer (AJCC) 7th edition, based on the following minimum workup:

  * Computed tomography (CT) chest/abdomen with contrast
  * Positron emission tomography (PET)/CT of the whole-body or skull base to mid-thigh
  * Patients must have regional adenopathy and have undergone endoscopic biopsy with endoscopic ultrasound (EUS)-proven peri-esophageal nodal involvement
* Subjects must have had no prior therapy for cancer of the esophagus
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* White blood cell count >= 3.0 K/cu mm
* Absolute neutrophil count >= 1.5 K/cu mm
* Platelets >= 100 K/cu mm
* Hemoglobin >= 8.0 g/dl (The use of transfusion or other invention to achieve Hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Serum ferritin < 2.0 X institutional upper limit of normal
* Woman of childbearing potential, a negative serum or urine pregnancy test
* Willingness to use adequate contraception for 12 months after completion of all therapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with cervical or Siewert 3 esophageal carcinoma, that are recommended by the multi-disciplinary tumor board to have treatment other than tri-modality chemo-radiation therapy (RT) followed by esophagectomy
* Subjects with AJCC 7th edition stage TxN0, T4b, and M1 disease
* Prior systemic chemotherapy for esophageal cancer; prior chemotherapy for another malignancy is allowable as long as it has been > 2 years since completion of therapy for previous malignancy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ferumoxytol or other agents used in the study
* Prior chest radiation or radiation for esophageal cancer
* History of other malignancy in the past 2 years except non-melanomatous skin cancer, breast ductal carcinoma in situ (DCIS) and low-risk prostate adenocarcinoma
* Medical contraindications to esophagectomy
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because chemoradiotherapy has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to the use of ferumoxytol as a contrast agent in the mother, breastfeeding should be discontinued if the mother receives ferumoxytol while nursing; men who are sexually active and not willing/able to use medically acceptable forms of contraception are also excluded from this study
* Subjects with multiple drug allergies and/or subjects who have had an allergic reaction to any intravenous iron replacement product or a known history of hypersensitivity to ferumoxytol
* Subjects with evidence of iron overload
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ferumoxytol
* Patients with renal insufficiency; glomerular filtration rate (GFR) < 60
* Adult patients who require monitored anesthesia for magnetic resonance imaging (MRI) scanning
* Subjects who have a contraindication for MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium (Gd) contrast material
* Subjects with known hepatic insufficiency or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Practical feasibility | Up to 18 weeks
  Will be assessed by successful accrual objectively, as a percentage of all subjects enrolled. Accrual success will be measured in binary fashion; successful accrual is considered a patient that enrolls and completes the entire trial. All other eligible patients will be considered an accrual failure. Practical feasibility will be considered a success if greater than 50%.
Technical feasibility of ultrasmall superparamagnetic iron oxide (USPIO) - magnetic resonance imaging (MRI) of the chest | Up to 18 weeks
  Will be evaluated in a descriptive manner. Image quality, readability (i.e. the ability for diagnostic radiologist to make an appropriate diagnostic conclusion, completion of ferumoxytol infusion, data acquisition, and completion of MR protocol.

SECONDARY OUTCOMES:
Accuracy of USPIO - MRI | Up to 18 weeks
  Accuracy, which is defined as the percentage of all patients or lymph nodes in which MRI with ferumoxytol correctly predicted the presence or absence of metastatic tumor, will be calculated.
Reason for accrual failure | Up to 18 weeks
  Descriptive statistical analysis of accrual failure will be conducted, counting the number of subjects who fail to complete the entire trial and the reasons for failure.
Report location and enhancement patterns on USPIO - MRI | Up to 18 weeks
Sensitivity and specificity of MRI imaging for all lymph nodes | Up to 18 weeks
  Sensitivities and specificities of ferumoxytol enhanced MRI prior to neoadjuvant chemoRT will be calculated using pathology finding as the gold standard. Each lymph node will be treated as an independent observation. The sensitivity and specificity will be compared with those from positron emission tomography (PET)/computed tomography (CT) findings using McNemar's test. Sensitivities and specificities of ferumoxytol enhanced MRI before surgery will also be calculated as a reference.
Sensitivity and specificity of PET/CT imaging | Up to 18 weeks
  Sensitivities and specificities of ferumoxytol enhanced MRI prior to neoadjuvant chemoRT will be calculated using pathology finding as the gold standard. Each lymph node will be treated as an independent observation. The sensitivity and specificity will be compared with those from PET/CT findings using McNemar's test. Sensitivities and specificities of ferumoxytol enhanced MRI before surgery will also be calculated as a reference.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Guimaraes, Principal Investigator — OHSU Knight Cancer Institute